CLINICAL TRIAL: NCT07407309
Title: Effects of Antenatal Delivery Room Visit and Companion Support During Labor on Maternal Comfort and Adaptation to Childbirth: A Randomized Controlled Trial
Brief Title: Antenatal Delivery Room Visit and Companion Support in Labor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nilgun Avci (Other)
Responsible Party: Sponsor-Investigator, Nilgun Avci, phD, Biruni University
Organization: Biruni University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Delivery Room Visit and Compan
Record Dates: First submitted 2026-02-06; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Pregnancy; Labor and Childbirth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Antenatal Delivery Room Visit and Companion Support (Experimental): Participants received an antenatal visit to the delivery room prior to labor and continuous companion support during the labor process, in addition to standard maternity care.
  Interventions: Behavioral: Antenatal Delivery Room Visit and Companion Support
- Control Group (No Intervention): Participants received standard maternity care without an antenatal delivery room visit and without continuous companion support during labor.

INTERVENTIONS:
Behavioral: Antenatal Delivery Room Visit and Companion Support — Participants received an antenatal visit to the delivery room prior to labor and continuous companion support during the labor process, in addition to standard maternity care.
  Arms: Antenatal Delivery Room Visit and Companion Support

SUMMARY:
This study evaluated whether an antenatal visit to the delivery room combined with companion support during labor improves comfort and adaptation to childbirth among pregnant women. The childbirth environment and lack of familiarity with the delivery room may increase anxiety and reduce comfort during labor. Supportive interventions before and during labor may help women adapt more positively to the childbirth process.

In this randomized controlled trial, pregnant women were assigned either to an intervention group that received an antenatal delivery room visit and continuous companion support during labor, or to a control group that received standard maternity care without these interventions. Maternal comfort and adaptation to childbirth were assessed using validated measurement tools after birth.

The results of this study aim to support evidence-based maternity care practices and highlight the importance of antenatal preparation and continuous support during labor to enhance women's childbirth experiences.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 years and older
* Gestational age between 24 and 40 weeks
* Planning a vaginal birth at the study hospital
* Able to communicate in Turkish
* Volunteered to participate and provided informed consent

Exclusion Criteria:

* High-risk pregnancy diagnosis
* Planned or emergency cesarean section
* Sensory or cognitive impairment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
Maternal Comfort During Childbirth | Within the first 2 hours after birth
  Maternal comfort assessed using the Childbirth Comfort Questionnaire.

SECONDARY OUTCOMES:
Adaptation to Childbirth (Midwife Assessment) | Within the first 2 hours after birth
  Adaptation to childbirth assessed by midwives using the Midwife Evaluation of Childbirth Adaptation Scale.

CONTACTS AND LOCATIONS:
Locations (1):
- State Obstetrics and Gynecology Hospital, Istanbul, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No